CLINICAL TRIAL: NCT02423798
Title: Accuracy and Performance Evaluation of the Medtronic New Generation Enlite Glucose Sensor in Conjunction With the Medtronic 640G System Components - in Clinic and at Home
Brief Title: New Generation Enlite Accuracy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Collaborators: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEP 296
Record Dates: First submitted 2015-03-23; First posted 2015-04-22 (Estimated); Results first posted 2017-09-25 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Diabetes
Keywords: Diabetes; Glucose sensor; Sensor accuracy and performance; CGM
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Open-label, single-sample design (Other): The trial has an open label design with a glucose sensor intervention. Only 1 sensor system is used in the trial (no comparator).
  As all subjects will receive identical devices and undergo the same experimental procedures, no randomization will be performed. Furthermore, neither subjects nor clinical staff will be blinded to the sensor readings, as knowing the sensor glucose readings will not affect the accuracy endpoint.
  Interventions: Device: Glucose sensor (Enlite)

INTERVENTIONS:
Device: Glucose sensor (Enlite) — This is a postmarket, interventional, open-label, non-randomized, single center clinical research trial. The trial will adopt a prospective single-sample design using the Yellow Spring Instruments (YSI) plasma glucose reference sampling procedure in the clinic and selfmonitoring of blood glucose (SMBG) plasma glucose reference sampling procedure at home. The trial will consist of 6 visits to the investigational site: a visit for informed consent procedures (Visit 0), a screening visit (Visit 1), 3 study visits (Visit 2-4) and a final examination (Visit 5).

SUMMARY:
The trial will investigate the accuracy and performance of a new sensor for continuous glucose monitoring (CGM), the (new generation) Enlite, CE-marked in 2013, in conjunction with the new Medtronic 640G system components.

To evaluate the accuracy and performance of the new generation Enlite sensor. This is a postmarket, interventional, open-label, non-randomized, single center clinical research trial.

The trial will adopt a prospective single-sample design using the Yellow Spring Instruments (YSI) plasma glucose reference sampling procedure in the clinic and self-monitoring of blood glucose (SMBG) plasma glucose reference sampling procedure at home.

DETAILED DESCRIPTION:
The trial will investigate the accuracy and performance (i.e. the life-time) of a new sensor for CGM, the (new generation) Enlite glucose sensor, CE-marked in 2013, in conjunction with the new Medtronic 640G system components. Accuracy and life-time of the sensor are important parameters contributing to the safety of patients and patient acceptance of this still fairly new technology.

The current trial investigates the accuracy of the new sensor in conjunction with the new 640G system components both in the clinic and at home. This enables us to assess the sensor accuracy in a well-controlled environment using a highly accurate laboratory glucose analyzer as reference as well as sensor accuracy during real-life conditions using a blood glucose meter as reference analyzer.

The data gathered in this trial will help to understand the effect of technological advancements made and can guide future development of glucose sensor for continuous glucose monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed the informed consent form prior to screening
* Age 18-74 years (both inclusive)
* Subject has been diagnosed with T1DM
* Subject is current insulin pump user for at least 3 months
* HbA1c 9.5%
* With the exception of T1DM, the subject is considered generally healthy upon completion of medical history, physical examination, vital signs, ECG and biochemical investigations as judged by the Investigator

Exclusion Criteria:

* Female of childbearing potential who is pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods (adequate contraceptive measures include sterilization, hormonal intrauterine devices, oral contraceptives, sexual abstinence, vasectomized partner)
* Subject has any condition that, in the opinion of the Investigator or qualified Investigational Centre staff, may preclude him/her from participating in the study and completing study related procedures.
* Subject has impaired vision or hearing problems that could compromise the handling of the device as determined by Investigator or qualified Investigational Centre staff
* Subject is unable to tolerate tape adhesive in the area of sensor placement
* Subject has any unresolved adverse skin condition in the area of sensor placement (e.g. psoriasis, rash, Staphylococcus infection)
* Subject has travel plans which would make it difficult for the subject to attend on-site study visits as scheduled
* Subject is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 30 days
* Subject known to be positive for Hepatitis B surface antigen (HBsAg) or Hepatitis C antibodies (or diagnosed with active hepatitis according to local practice).
* Positive result to the screening test for HIV-1 antibodies, HIV-2 antibodies or HIV-1 antigen according to locally used diagnostic testing
* Significant history of alcoholism or drug/chemical abuse as per investigator's judgment, current regular alcohol consumption of more than 1 unit per day for women and more than 2 units per day for men [1 unit of alcohol equals 1 beer (330 mL), 1 glass of wine (120 mL), or 1 glass of spirits (40 mL)], or a positive result in the urine drug/alcohol screen at the screening visit

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All Subjects
Pre-assignment Details: All Subjects
Groups:
- All Subjects: All subjects will receive identical devices and undergo the same experimental procedures.
Period: Overall Study
Arm/Group | All Subjects
Started | 24
Completed | 21
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- All Subjects: All Subjects
Arm/Group | All Subjects
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.6 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Region of Enrollment [Count of Participants; unit: Participants]
  Europe | 24

OUTCOME MEASURES:

1. Primary Outcome: Sensor Accuracy
Description: Sensor values were compared to YSI plasma glucose values, which is considered as the gold standard, during the frequent sample testing day (day 3). MARD = Mean of ((Absolute difference of YSI reference and Sensor glucose values / YSI reference glucose values) * 100).
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | All Subjects
Number analyzed (Participants) | 24
percentage | 9.13 (7.14)
Statistical Analysis 1: Comparison: All Subjects; Test type: Other; Mean = 9.13

2. Primary Outcome: Consensus Error Grid Analysis of Paired Sensor and Reference Plasma Glucose Values
Description: All analysis performed using the Consensus Error Grid (or Parkes error grid) comparing the paired sensor and YSI reference glucose values.
  Zone A is defined in the Parkes error grid as the zone of "clinical accurate measurements with no effect on clinical action." Zone B as "altered clinical action with little or no effect on clinical outcome.". Ideal situation is 100% in Zone A + B.
Time Frame: 4 months
Measure: Number; unit: percentage
Arm/Group | All Subjects
Number analyzed (Participants) | 24
percentage | 100.0

3. Primary Outcome: Sensor Survival
Description: sensor survival in hours
Time Frame: 4 months
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | All Subjects
Number analyzed (Participants) | 24
hours | 130.8 [115.7 to 145.9]

ADVERSE EVENTS:
Arm/Group | All Subjects
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 5/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Subjects (N=24)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
itching at sensor insertion (General disorders) | 2 (2)
hematoma at insertion (General disorders) | 1 (1)
erythema at insertion site (General disorders) | 1 (1)
mild erythema (Skin and subcutaneous tissue disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days